CLINICAL TRIAL: NCT01036971
Title: Screening Protocol for the Evaluation of Potential Research Subjects
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999906415; 06-DA-N415
Record Dates: First submitted 2009-12-18; First posted 2009-12-21 (Estimated); Last update posted 2026-01-28 (Actual); Status verified 2025-12-17

CONDITIONS: Addiction
Keywords: Physical Examination; Medical Information; Assessment; Blood Work; Screening
MeSH Terms: conditions — Behavior, Addictive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: potential research subjects

SUMMARY:
Background:

- The Neuroimaging Research Branch of the National Institute on Drug Abuse (NIDA) is interested in developing a pool of potential research participants who may be eligible for research studies on drug abuse and addiction, pharmacological and psychosocial therapies for substance addiction, and the long-term effects of drugs on the development, function, and structure of the brain and other organ systems. To develop this pool of potential participants, researchers intend to screen adolescents and adults who may be eligible for future research studies.

Objectives:

- To identify, recruit, and screen participants for NIDA neuroimaging research protocols.

Eligibility:

- Individuals 18 years of age and older who are able to provide informed consent.

Design:

* Eligible participants will undergo two screening interviews: a telephone interview and an in-person interview. The phone interview will determine eligibility for the in-person interview. Adolescents who are eligible for further screening must bring a parent or guardian with them to the in-person interview.
* The in-person interview may require up to five visits to the NIDA clinical center. The in-person visit will involve any or all of the following procedures: (1) full physical examination and medical history; (2) psychiatric interview; (3) psychological testing; (4) electrocardiogram; (5) samples of blood, urine, and hair; and (6) other minimally invasive procedures as directed by the research staff.
* During the screening process, participants will be explicitly asked for permission to recontact them after the 1-year duration of the screening protocol. For minors, both the adolescent and the parent/guardian must agree to future contact.
* No clinical care will be provided under this protocol.

DETAILED DESCRIPTION:
This protocol describes the screening process used by the National Institute on Drug Abuse (NIDA IRP) to assess potential research participants' eligibility for entering protocols of the NIDA/IRP. Through its clinical research protocols, the IRP attempts to: elucidate the nature of drug abuse and addiction; determine the potential use of new therapies, both pharmacological and psychosocial; and decipher the long-term effects of drugs of abuse on the development, maturation, function, and structure of the brain and other organ systems. In support of the IRP's' work, the scientific goal of this screening protocol is to assess potential research participants' eligibility for the IRP's research studies. Screening will include medical and psychological tests and procedures. The data collected during screening are a unique and valuable source of information that aids in the IRP's mission. Therefore, a secondary goal of this protocol is to obtain data that characterizes the population of subjects contacting the IRP about research participation and to analyze data so obtained, such as that on the prevalence and co-occurrence of pregnancy, HIV/AIDS, viral hepatitis, and related diseases. The population screened includes male and female adults age >= 18. Screening procedures include standard medical and psychological tests and procedures are minimal risk. There is no direct benefit to subjects. Participants are paid for undergoing the screening process.

Most genetics data will be collected under the aegis of other protocols and will be compared with data collected under this study. Some studies require genotyping to be done as part of screening. Those DNA samples will be stored so that if active or returning participants are screened for future studies requiring genotyping during screening an additional blood draw will not be required.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Males and females ages 18 or older.

EXCLUSION CRITERIA:

1. Phone screen: Subjects who are unable to understand or adequately answer questions posed in the phone screen.
2. Phone screen and in-person screen: Subjects unable to provide informed consent.
3. Pregnant women

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Screening protocol for all NIDA clinical studies
Sampling Method: Non-Probability Sample
Enrollment: 6967 (Actual)
Dates: Start 2006-08-23 (Actual)

PRIMARY OUTCOMES:
Screening for NIDA studies | baseline
  Screening for NIDA studies

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Leggio, M.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Biomedical Research Center (BRC), Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
No plan depicted in protocol.